CLINICAL TRIAL: NCT03443791
Title: Cytomegalovirus (CMV) Vaccines: Reinfection and Antigenic Variation
Acronym: CMV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, William J. Britt, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-010810006
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Cmv Congenital; CMV Viremia
Keywords: CMV; Congenital Birth; Infectious Diseases
MeSH Terms: conditions — Cytomegalovirus Infections; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women enrolled (Experimental): pregnant women enrolled in trial
  Interventions: Diagnostic Test: Women Enrolled
- newborns of female study participants (Other): newborns will be tested to determine if virus is present.
  Interventions: Diagnostic Test: Newborns of Female Study Participants

INTERVENTIONS:
Diagnostic Test: Women Enrolled — Diagnostic Testing will be performed. Results of individual test results will determine the degree of intervention offered.
  Arms: women enrolled
Diagnostic Test: Newborns of Female Study Participants — Newborns will be tested after birth as soon as possible for CMV positivity.
  Arms: newborns of female study participants

SUMMARY:
The objectives of the protocol are to determine if a structured cognitive-behavioral interventional counseling of pregnant women can limit acquisition of human cytomegalovirus (HCMV) during pregnancy that we believe, will in turn decrease the incidence of congenital HCMV infections in this highly seroimmune population. Previously, investigators have demonstrated the success of a similar approach in pregnant women without previous evidence of HCMV infection (non-immune women) but to date, there is no evidence that such an approach will alter the incidence of congenital HCMV infections in seroimmune women. This protocol will take advantage of recently derived data in this maternal population that has identified sources HCMV exposure in women in this population and thus provided new insight into targeted counseling interventions that could limit maternal acquisition of HCMV. The primary endpoints of this study will be a 50% reduction in the overall incidence of congenital HCMV infections in this maternal population with secondary endpoints being efficient uptake of behavioral recommendations and modifications of simple hygiene behaviors that have previously been shown to decrease exposure and acquisition of HCMV.

DETAILED DESCRIPTION:
The proposed cognitive-behavioral intervention protocol to modify the risk of exposure and acquisition of HCMV in pregnant women will include a two components. The first component of the trial will consist of a pilot study in which 100 women enrolled in the parent study will be asked to participate in this substudy. We will target women with young children in the household and households with more than 5 inhabitants as these two characteristics have been shown to be associated with virus excretion in pregnant women in this population, and by inference, exposure and acquisition of HCMV during pregnancy in this maternal population. Women will be counseled at enrollment utilizing both a brief counseling session that will provide basic information about HCMV and congenital HCMV (cCMV) infections, and an individualized behavioral skills session. A take home packet describing the; (i) cCMV infections, (ii) routes of virus acquisition/spread and measures to limit virus spread, and (iii) guidance in behavior modifications to reduce risk of exposures and infection with HCMV will be provided. Enrollees will be seen during their following prenatal visits and asked to complete a questionnaire that will include a self-assessment of adherence to recommended risk reduction behaviors, understanding of routes of HCMV transmission, and importantly, the burden of introducing recommended risk reduction practices into their daily routines. In addition, we will poll these women on the most effective components of the cognitive-behavioral intervention pilot. Data derived from these questionnaires will represent the outcome of this pilot study and will permit us to modify the strategy that will be deployed in the larger intervention trial.

The second component will consist of a larger trial of cognitive-behavioral intervention trial to limit HCMV exposure and acquisition in pregnant women in this maternal population. Women \ will complete a standard questionnaire that will provide demographics such as description of housing, number of people in household, number and ages of children. Information will also be gathered on number and age of sexual partners, previous STIs, and if partner currently resides in household. Standard of care counseling will include discussion of sources of infections and routes of acquisition. After enrollment, women will be randomized to standard of care of counseling or the HCMV exposure risk reduction intervention strategy by assignment of every other enrollee to the intervention cohort. Women enrolled in the exposure risk reduction intervention will receive standard of care and receive an individualized behavioral skills session from a trained nurse or health educator (see following section). As part of enrollment in this study, all women will provide permission to screen their newborn infants or any specimens from miscarriages or fetal loss for HCMV infection. Samples of prenatal blood specimens collected as part of routine care will be stored for future use and enrollment saliva swab, vaginal swab, and urine will be obtained and stored for studies of viral load and baseline viral genomic diversity. The behavioral intervention group will also watch a short video detailing basic information about HCMV, the natural history of HCMV infections (sources and routes of transmission), and consequences of maternal infection during pregnancy to the outcomes of pregnancy. Within this video will be explicit and specific descriptions of exposures, such as kissing young children on the mouth, handling objects that have been or could have been in the mouths of young children, and the importance of hygiene after exposure to urine during diaper changing. After viewing the video, a nurse (or health educator) specifically trained to reinforce the information in the video will provide a brief behavioral skills session, and distribute a take home packet containing an information pamphlet. Study participants will receive weekly brief text messages for the initial 12 weeks to deliver reminders of recommended behaviors to limit risks of exposures. To power this study for a 50% difference in the outcome of pregnancy (delivery of a infant with cCMV infection) in a population with the incidence of cCMV of 0.6%, we have estimated that 4300 women will be required. Between the two hospitals and clinics that serve the population in this study, approximately 4700 deliveries take place per year. Our plan is to enroll patients over 2 years, thus we believe that we can enroll 5,000 women in this study.

ELIGIBILITY:
Inclusion:

* Women in Ribeirao Preto who receive maternity care through the Hospital Das Clinicas, University of São Paulo and the Mater Hospital
* enrollment in prenatal care before 23 weeks gestation

Exclusion:

* late enrollment in prenatal care, after 23 weeks gestation
* known major fetal anomalies or demise
* planned termination of pregnancy
* intention of the patient to deliver at a non-study hospital
* referral for high risk prenatal care

Ages: 1 Hour to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
A 50% reduction in the overall incidence of congenital HCMV infections in this maternal population | baseline through 60 months
  Participants will be tested using urine and blood to determine positivity for CMV

SECONDARY OUTCOMES:
efficient uptake of behavioral recommendations and modifications of simple hygiene behaviors | baseline through 60 months
  Participants are educated on personal hygiene behaviors which have previously been shown to decrease exposure and acquisition of HCMV. Study visits will included survey for these questions.

CONTACTS AND LOCATIONS:
Overall Officials: William J. Britt, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Sao Paulo, São Paulo, Brazil